CLINICAL TRIAL: NCT00523029
Title: Self-Management of Depression and Medical Illness
Brief Title: Developing a Self-Management Program for People With Depression and Chronic Medical Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Isabel T. Lagomasino, MD, MSHS, Study Principal Investigator, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R34MH072631 (NIH); R34MH072631 (NIH); DSIR 82-SEPC
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Depression
Keywords: Self-management programs; Chronic medical illness
MeSH Terms: conditions — Depression

ARMS (1):
- 1 (Experimental): Participants will receive a chronic disease self-management program
  Interventions: Behavioral: Chronic Disease Self-Management Program

INTERVENTIONS:
Behavioral: Chronic Disease Self-Management Program — Chronic disease self-management is a 6-week group program that teaches participants how to manage their chronic medical illness. Group leaders, also suffering from a chronic medical condition, will lead discussions based on the following topics: nutrition; exercise; appropriate use of medications; ways to communicate effectively with family, friends, and health care professionals; and how to make informed treatment decisions.

SUMMARY:
This study seeks to adapt an existing chronic disease self-management program for people with both chronic medical illness and depression.

DETAILED DESCRIPTION:
Depression is a common but serious disorder that affects millions of people every year. Depression can severely impact people's lives, causing them to often feel sad and hopeless as well as affecting their sleep patterns, concentration, and energy levels. Treatment typically includes a combination of antidepressant medication and talk therapy. This study will evaluate the effectiveness of an adapted group education program typically used for chronic medical illness in improving the health status, health behaviors, and use of health care services among people with depression and a chronic illness.

Participants in this open-label study will attend a group education program used to manage chronic medical illness. Group sessions will be held for 2.5 hours, once a week, for 6 weeks. Group leaders, also suffering from a chronic medical condition, will lead discussions based on the following topics: nutrition; exercise; appropriate use of medications; ways to communicate effectively with family, friends, and health care professionals; and how to make informed treatment decisions. Participants will also complete two surveys: one at the beginning of the study and one at the end. The first survey will ask basic questions related to participants' health status and any feelings of stress, anxiety, or sadness. The second survey will include a brief interview that will require participants to describe their experience in the group sessions and to suggest ways of improving the program to better accommodate people with depression and chronic illness. Responses to questions will be used to enhance the effectiveness of the group education program for treating people with both depression and a chronic medical condition.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Currently attending the Edward R. Roybal Comprehensive Health Center or the LAC+USC Outpatient Department for primary care
* English- or Spanish-speaking
* Screens positive for major depressive disorder or minor depression based on the PRIME MD PHQ-9
* Suffers from a chronic medical illness (e.g., lung disease, asthma, emphysema or trouble breathing; heart disease or heart problems; high blood sugar or diabetes; arthritis or rheumatism)

Inclusion Criteria for Group Leaders:

* Prior experience facilitating a chronic disease self-management program within 6 to 9 months of study entry (including the groups held at Roybal Comprehensive Health Center)

Exclusion Criteria for Patients:

* Acutely suicidal
* Screens positive for bipolar disorder, psychotic disorder, or cognitive impairment disorder
* History of alcohol or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2006-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
PRIME-MD Patient Health Questionnaire (PHQ-9) | Measured at Week 8
Qualitative interviews of participants and leaders | Measured at Week 8
Post-intervention assessments, including self-efficacy, health behaviors, health status, and service utilization | Measured at Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Isabel T. Lagomasino, MD, MSHS, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Edward R. Roybal Comprehensive Health Center, Los Angeles, California
  - LAC and USC Medical Center, Outpatient Department, Los Angeles, California